CLINICAL TRIAL: NCT04120909
Title: MARC-2: MARKERS AND RESPONSE TO CRT in Non-LBBB
Acronym: MARC-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Kevin Vernooy, dr. Kevin Vernooy, Maastricht University Medical Center
Other Study IDs: 2018-0863
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Cardiac Resynchronization Therapy, Non-LBBB, QRS Area
Keywords: cardiac resynchronization therapy, non-LBBB, QRS area
MeSH Terms: interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cardiac resynchronization therapy — Biventricular pacing according to current standards.

SUMMARY:
The purpose of the MARC-2 study is to investigate the relation of the QRS area, determined by vectorcardiography, and response to Cardiac Resynchronization Therapy (CRT) in patients with a wide QRS complex and without a typical left bundle branch block; the interrelationship as well as the potential predictive power of this biomarker, as well as other clinical biomarkers on a hierarchal composite endpoint (death, heart failure hospitalizations, heart failure complaints and cardiac function) will be evaluated.

The main biomarker that is studied is the QRS area, but also other electrocardiographic, echocardiographic markers, blood markers and clinical markers will be studied.

DETAILED DESCRIPTION:
For the purpose described in the brief summary, the MARC-2 study investigators have set an aim of including 800 patients in 2 inclusion years, in 30 centres accross Europe and Israel. Inclusion will be general patients indicated for (de novo or upgrade) implantation a (Medtronic) CRT-pacemaker or -ICD, as according to current ESC heart failure guidelines. Exclusion criteria are, age below 18 years, (planning) childbearing, baseline > 5% RV-pacing, listing for transplantation or inotropic dependency, structural heart disease for which invasive therapy is pending, or inability/unwillingness to sign written informed consent. All QRS morphologies, with duration >/= 130ms are included because multiple LBBB definitions exist and excluding patients on one definition will leave room for questions about the definitions used. (Bio)markers that are collected are electrocardiographic/vectorcardiographic/echocardiographic/blood-/CMR/ and device-based parameters that have shown prior association to outcomes in CRT, with special attention to vectorcardiographic QRS area. The primary endpoint will be a hierarchal (Packer) score of collected heart failure related endpoints including death/LVAD/cardiac transpland/heart failure hospitalizations/echocardiographic remodelling and NYHA improvement. Follow-up for clinical endpoints will be 12 months; with echocardiographic follow-up at 6 months. Clinical endpoints are subject to adjudication committee assessment. Core-labs exist to assess electrocardiographic, echocardiographic and CMR-data.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to be implanted with a CRT-pacemaker or CRT-defibrillator
* Subject has NYHA class I, II, III or ambulant IV
* Subject has LV dysfunction (LVEF</=35%)
* Subject is in sinus rhythm on an ECG less than 45 days before CRT implantation
* Intrinsic QRS duration is >/=130ms (of either QRS morphology) within 30 days prior to CRT device implantation
* Subject receives optimal heart failure oral medical therapy (ACE inhibitor and/or ARB and Beta Blockers), and is on a stable medication scheme for at least 1 month prior to enrolment
* Subject is willing to sign informed consent form
* Subject is 18 years or older

Exclusion Criteria:

* Subject has a pacemaker/ICD with >5% RV pacing.
* Subject receives CRT-D replacement or is upgraded from CRT-P to CRT-D
* Subject experienced a recent myocardial infarction, within 40 days prior to enrollment
* Subject underwent coronary artery bypass graft (CABG) or valve surgery, within 90 days prior to enrollment
* Subject is post heart transplantation, or is actively listed on the transplantation list, or has reasonable probability (per investigator's discretion) of undergoing transplantation in the next year
* Subject is implanted with a left ventricular assist device (LVAD), or has reasonable probability (per investigator's discretion) of receiving a LVAD in the next year
* Subject is on continuous or uninterrupted infusion (inotropic) therapy for heart failure
* Subject has permanent 2nd or 3rd degree AV-block
* Subject has severe aortic stenosis (with a valve area of <1.0 cm2 or significant valve disease expected to be operated within study period)
* Subject has complex and uncorrected congenital heart disease
* Subject has a mechanical right heart valve
* Subject has a life expectancy of less than one year in the opinion of the investigator
* Pregnant or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth control
* Subject is enrolled in one or more concurrent studies that would confound the results of this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study group to be recruited will consist of heart failure patients (NYHA I-IV), male and female, with a reduced left ventricular ejection fraction (LVEF</=35%) and ventricular dyssynchrony (QRS>/=130ms) as measured prior to implantation of a CRT device. Each study subject receives a CRT device with a class I or II indication according to the current CRT ESC/AHA guidelines.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
CRT response score will assess patient improvement including all-cause mortality, heart failure hospitalization, LVESVi reduction, and NYHA class improvement | 12 months
  Hierarchical endpoint based upon the concepts presented by Packer (Packer, Circulation 2016)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Stipdonk AMW, Ter Horst I, Kloosterman M, Engels EB, Rienstra M, Crijns HJGM, Vos MA, van Gelder IC, Prinzen FW, Meine M, Maass AH, Vernooy K. QRS Area Is a Strong Determinant of Outcome in Cardiac Resynchronization Therapy. Circ Arrhythm Electrophysiol. 2018 Dec;11(12):e006497. doi: 10.1161/CIRCEP.118.006497. PMID 30541356